CLINICAL TRIAL: NCT00643123
Title: A Double-Blind, Placebo Controlled Augmentation Study With Allopurinol for Treatment Resistant Mania
Brief Title: Allopurinol Add-on Treatment for Refractory Mania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Itai Danovitch, Chairman, Department of Psychiatry, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB8981
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Bipolar Disorder; Mixed Mania; Treatment-Resistant Mania
Keywords: Bipolar Disorder; Mania; Mixed mania; Allopurinol; Treatment-Resistant mania
MeSH Terms: conditions — Bipolar Disorder; Mania | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Allopurinol (Experimental): Subjects will be randomized to allopurinol at a fixed dose of 300 mg/day for the first week and then 600mg/day while continuing their current medications during the 7-week study. A battery of assessments will be administered at baseline and weeks 1, 2, 4, 6 after baseline. At each assessment, subjects will also be asked about side effects including potential side effects of allopurinol. Side effects will be assessed by the Treatment Emergent Side Effects Scale. Serum levels of lithium, valproic acid, carbamazepine, atypical antipsychotics or atypical antipsychotic metabolite, uric acid blood levels will be drawn at screen and at week 6 after baseline. Subjects taking only lithium, valproic acid, and/or carbamazepine will also have their serum levels drawn at week 2.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator): Subjects will be randomized to placebo and will follow the same protocol as the allopurinol group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Allopurinol — 300-600 mg/day over a 6 week period
  Other Names: Zyloprim
  Arms: Allopurinol
Other: Placebo — Inactive substance
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy of allopurinol as an augmentation agent for treatment resistant mania and mixed mania.

DETAILED DESCRIPTION:
Bipolar disorder is a severe mental disorder with episodes of mania and depression. Current medications for mania can have significant side effects, high costs and the need for blood monitoring. The purpose of this research study is to study the effectiveness of allopurinol, in combination with lithium or valproic acid or carbamazepine, for treatment-resistant bipolar mania and mixed mania. This research study is designed to test the safety and/or effectiveness of allopurinol that has been approved by the U.S. Food and Drug Administration (FDA) for recurrent calcium renal calculus, gout, hyperuricemia (cancer and tumor lysis syndrome), but it is not approved for use in treatment-resistant bipolar mania or mixed mania.

Participants in this double-blind study will be randomly assigned to one of two study groups. The first group will receive the study medication of allopurinol while the second group will receive a placebo. These will be taken in conjunction with current medications and doses. The study will last for 7 weeks (an initial screening, a baseline visit and 4 follow-up visits at weeks 1,2,4, and 6). The initial screening visit will be used to determine whether or not the subject is able to participate in the study. The following will be conducted during the screening visit: Review of medical and psychiatric history along with standard psychiatric assessment exams; Physical examination, including review of prior and current medications and adverse drug effects; An electrocardiogram (ECG) - a painless test which is done by attaching straps or pads to your limbs and chest and recording the electrical pattern of your heart, will be done to record your heart rhythm; About 5 tablespoons of blood will be drawn to assess basic laboratory values that show if you are healthy enough to participate in the study; Blood levels of lithium, valproic acid, and/or carbamazepine will be measured; A urine sample will be collected to test for the presence of illegal drugs and for pregnancy test (if you are a female of child-bearing potential); Collection of demographic data (e.g., age, gender, marital status, social and vocational status) and other information including health beliefs, and knowledge of illness. At the baseline visit the participant will be given questionnaires related to mood, quality of life, disability, medications, and side effects. The participant's vitals (temperature, weight, heart rate, and blood pressure) will be measured. The participant will be randomized to treatment (300 mg of allopurinol/day) or placebo. After week one at the Week 1 visit, those that have tolerated the dosage of allopurinol will get an increased dosage. The participant will also complete a set of questionnaires. Vitals will be taken. The remaining follow-up visits will be similar to visit one except that there will be no more increases in dosage; Week 2 will include a blood draw to measure levels of lithium, valproic acid, and/or carbamazepine in the participant's blood, and the final visit at Week 6 will in addition include a blood draw, and exit physical exam, and a urine sample will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between ages 18 and 70.
* Subjects must meet DSM-IV criteria for bipolar disorder, most recent episode manic or mixed, at the time of screening confirmed by the Mini International Neuropsychiatric Interview (MINI).
* Subjects must be taking at least one medication for mania (lithium, valproic acid, carbamazepine) at a therapeutic dose for at least 4 weeks.
* Subjects must have non-response or partial response to medications as evidenced by Young Mania Rating Scale (YMRS) score greater than or equal to 14 at screening and at baseline.
* Female subjects must be either postmenopausal for at least 1 year, surgically sterile, abstinent or practicing an effective method of birth control if sexually active. Female subjects must also have a negative urine pregnancy test at screening, baseline and other time points throughout the study.
* Subjects must be able and willing to comply with self-administration of medication or have consistent help/support available.
* Subjects must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Subjects must be able and willing to meet or perform study requirements (e.g. answer self-administered questionnaires).
* Subjects must be willing to allow study staff to contact subject's regular psychiatrist while the subject is in the study.

Exclusion Criteria:

* Subjects who are unable to provide informed consent.
* Subjects with a serious, unstable medical illness (such as cardiovascular, respiratory, neurologic, hematologic, renal, hepatic, endocrine, immunologic, or other systemic illness), a history of cerebrovascular disease, uncontrolled diabetes mellitus or AIDS. Subjects with chronic illness must be stable and otherwise physically healthy on the basis of a physical examination, medical history, electrocardiogram and the results of blood biochemistry, hematology tests and a urinalysis.
* Subjects with a history of substance abuse or dependence (excluding nicotine and caffeine) according to DSM-IV criteria within last 4 weeks.
* Subjects taking azathioprine, mercaptopurine, apalcillin, and/or amoxicillin.
* Subjects taking dopamine agonists and/or anti-psychotics.
* Subjects who have been intoxicated with alcohol or illicit drugs within 3 days prior to baseline.
* Subjects with a history of severe pre-existing gastrointestinal narrowing or inability to swallow oral study medication whole with the aid of water.
* Female subjects who are pregnant or nursing.
* Subjects who have previously participated in this study.
* Subjects with an anticipated life expectancy of 6 months or less.
* Subjects who have received an experimental drug or used an experimental medical device within 1 month of screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Danovitch, M.D., Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Fan A, Berg A, Bresee C, Glassman LH, Rapaport MH. Allopurinol augmentation in the outpatient treatment of bipolar mania: a pilot study. Bipolar Disord. 2012 Mar;14(2):206-10. doi: 10.1111/j.1399-5618.2012.01001.x. PMID 22420596

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 8 subjects screen failed; 5 subjects did not qualify at Baseline. 13 total subjects were not randomized
Period: Overall Study
Arm/Group | Allopurinol | Placebo
Started | 15 | 12
Completed | 10 | 11
Not Completed | 5 | 1
Not completed — Lost to Follow-up | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allopurinol | Placebo | Total
Number analyzed (Participants) | 15 | 12 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race or Ethnicity: Caucasian | 9 | 8 | 17
  Race or Ethnicity: African-American | 3 | 4 | 7
  Race or Ethnicity: Hispanic | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 15 | 12 | 27
Marital Status [Count of Participants; unit: Participants]
  Never Married | 8 | 6 | 14
  Married | 1 | 3 | 4
  Divorced | 4 | 3 | 7
  Not Reported | 2 | 0 | 2
Employment Status [Count of Participants; unit: Participants]
  Employed | 4 | 4 | 8
  Unemployed | 9 | 6 | 15
  Disabled | 1 | 2 | 3
  Student | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Young Mania Rating Scale (YMRS)
Description: The YMRS is an 11-item, clinician-administered rating scale to assess the severity of manic symptoms before, during and after treatment. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. A score of 0 indicates the behavior is absent, whereas a score of 4 or 8 indicates the behavior is present and severe.
  The change in score between Baseline and the Completion Visit will be reported. Ideally, the two time points will be Baseline and 6 Weeks after Baseline, but, if a subject terminates early, his/her last YMRS score will be carried forward to the final visit.
  The scores from each question are added together to form a total score ranging from 0 to 60, with higher scores indicating a greater severity of symptoms. A score of 0-12 indicates the absence of mania or a very mild manic state, a score of 13-20 or higher indicates a mild man
Time Frame: 7 weeks (Baseline and 6 weeks (or last visit date) after baseline
Population: 27 subjects were randomized but 4 (3 from the Treatment group and 1 from the Control group) withdrew from the study immediately following the baseline visit. Therefore, a second time point was unavailable for these subjects.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 12 | 11
units on a scale | -12.3 (1.9) | -9.6 (2.7)
Statistical Analysis 1: Comparison: Allopurinol vs Placebo; Test type: Other; p = .45, t-test, 2 sided; Mean Difference (Final Values) = 2.9, Standard Error of Mean 2.3

2. Secondary Outcome: Hamilton Depression Scale (HAM-D)
Description: The Hamilton Depression Rating Scale (HAM-D) is a clinician-administered tool used to determine a patient's level of depression before, during, and after treatment. A 28-item HAM-D form was used but only the first 17 questions are used in the assessment for depression. Of the first 17 questions, eight items are scored on a 5-point scale, ranging from 0 = not present to 4 = severe. Nine are scored from 0-2. The sum of the scores from the first 17 questions is: 0-7 = normal, 8-13 = mild depression, 14-18 = moderate depression, 19-22=severe depression and ≥ 23=very severe depression.
  Questions 18-28 are scored similarly and assess sleep disorders, paranoid behavior, motor dysfunction, psychosis, and weight gain, etc.
Time Frame: 7 weeks
Population: No data displayed because no data was collected prior to closing of the research unit.
Arm/Group | Allopurinol | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Placebo | Allopurinol
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 1/12 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | Allopurinol (N=15)
Suicidal thoughts and plan (Psychiatric disorders) | 0 (0) | 1 (1)
Medication non-compliance (Psychiatric disorders) | 0 (0) | 1 (1)
Inflamed prostate (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Subject complained about enlarged prostate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes